CLINICAL TRIAL: NCT01765725
Title: Coping With Chronic Fatigue Syndrome: Development of a Community-based Patient Education Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Stiftelsen Helse og Rehabilitering (Other)
Responsible Party: Principal Investigator, Unni Sveen, Associate professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2011/894/REK nord; 2011/894/REK nord (Registry Identifier: REK nord); 36IAJ3 (Other Grant/Funding Number: Extra Stiftelsen Helse og Rehabilitering)
Record Dates: First submitted 2013-01-04; First posted 2013-01-10 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Chronic Fatigue Syndrome; Coping; Patient Education
Keywords: Chronic Fatigue Syndrome; Coping; Patient education
MeSH Terms: conditions — Fatigue Syndrome, Chronic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control group (No Intervention): The control group will be offered to take part in the patient education group as soon as they have completed the last outcome evaluations
- Patient education program (Experimental): Patient education program
  Interventions: Behavioral: Patient education program

INTERVENTIONS:
Behavioral: Patient education program — Patient education program, 8 meetings, every other week, 2,5 hours per meeting.
  Arms: Patient education program

SUMMARY:
The aim of the study is to develop, carry out, evaluate and measure the effects of a new patient education program for patients with Chronic Fatigue Syndrome (CFS)in primary healthcare.

In an randomized controlled trial design the effects of the patient education program on coping, physical functioning, fatigue, pain, acceptance, anxiety, depression, quality of life, self- efficacy, and illness perception will be compared with treatment as usual.

The results of the main project will lead to the elaboration of the final patient education program that can be implemented in primary health care, as well as development of a training program for future program-conductors.

DETAILED DESCRIPTION:
The project is a single blind randomized controlled trial. A total of 150 participants will be included in this study and randomly allocated to the intervention- or the control group. The 75 participants in the intervention group will be allocated to 6 groups. The control group will be offered to take part in the patient education program as soon as they have completed the last outcome evaluations.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Meets Fukuda's research diagnostic criteria and Canadian CFS case definition
* Has given oral and written informed consent
* Able to tak part in the program that lasts 2,5 hours in addition to transport to and from the location for intervention.

Exclusion Criteria:

* Psychosis or other severe psychiatric diseases, severe personality disturbances and/or substance dependency
* Pregnancy
* Not being able to understand, speak and read Norwegian
* Not willing to accept random assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2011-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
SF-36, subscale Physical functioning. | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in physical functioning.
Illness Management Questionnaire (IMQ). | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in ways of coping with CFS.

SECONDARY OUTCOMES:
The SF-36 (total score and subscale role limitations due to physical limitations). | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  The SF-36 total score measures change in functional status related to health. The subscale measures change in role limitations due to physical limitations.
Fatigue Severity Scale (FSS). | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in fatigue-related severity, symptomatology, and functional disability.
Illness Cognition Questionnaire (ICQ) | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measure change in helplessness, acceptance, and perceived benefits.
The Fennell Phase Inventory (FPI) | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in coping and progression through four phases: crisis phase, stabilization phase, resolution phase, and integration phase.
Hospital Anxiety and Depression Scale (HADS) | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in anxiety and depression.
Perceived Stress Scale (PSS)- 10 items | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in global perceived stress.
Brief Illness Perception Questionnaire (BIPQ) | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in cognitive and emotional representations of illness.
Self-efficacy Scale (SE24) | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in perceived control with respect to CFS complains.
Self-defined fatigue and pain scale | T0: Baseline, T1: After 4 months, T2: After 10 months, T3: After 16 months.
  Measures change in perceived fatigue and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Unni Sveen, Ph.d., Study Director — Oslo University Hospital; Irma Pinxsterhuis, M.Sc., Principal Investigator — Oslo University Hospital; Dag Kvale, Ph.d., Study Chair — Oslo University Hospital
Locations (1):
- Irma Pinxsterhuis, Oslo, Norway